CLINICAL TRIAL: NCT00282360
Title: Effect of Metabolic Therapy in Patients With Chronic Ischemic Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SR05-1-5
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2006-01-26 (Estimated); Status verified 2004-05

CONDITIONS: Coronary Artery Disease; Type II Diabetes Mellitus
Keywords: coronary artery disease; diabetes mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine

SUMMARY:
Patients with coronary artery disease have an abnormal cardiac metabolism. The hypothesis of this study is that shifting cardiac metabolism from free fatty acids to glucose will improve myocardial ischemia

DETAILED DESCRIPTION:
The present study will evaluate the effect of free fatty acid inhibition with Trimetazidine on silent myocardial ischemia and total ischemic burden in coronary artery disease patients with type II diabetes.

Patients will undergo ambulatory ECG monitoring at baseline and will be randomized to receive on top of thei standard anti-anginal therapy trimetazidine or placebo for 6 months. Patients will repeat the ambulatory ECG monitoring at the end of the study

ELIGIBILITY:
Inclusion Criteria:

coronary artery disease type II diabetes mellitus -

Exclusion Criteria:

unstable coronary artery syndromes impaired liver and kidney function

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-02; Study Completion 2003-10

PRIMARY OUTCOMES:
total ischemic burden
silent ischemia

SECONDARY OUTCOMES:
symptomatic myocardial ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Marazzi, MD, Principal Investigator — H San Raffaele EUR